CLINICAL TRIAL: NCT07036809
Title: Assessment of Antithrombin III, Protein C, Protein S and D-dimer in Acute Leukemia
Status: Completed | Type: Observational
Sponsor: Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy (Other)
Responsible Party: Sponsor-Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Organization: Al-Azhar University (Other)
Other Study IDs: clinicalpath1
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemia
Keywords: acute leukemia; Antithrombin III; protein C; Protein S; D Dimer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- acute lymphoblastic leukemia: patients diagnosed with acute lymphoblastic leukemia.
  Interventions: Diagnostic Test: Antithrombin III; Diagnostic Test: Protein C; Diagnostic Test: Protein S; Diagnostic Test: D-dimer; Diagnostic Test: Flow cytometry immunophenotyping
- acute myeloid leukemia: patients diagnosed with acute myeloid leukemia.
  Interventions: Diagnostic Test: Antithrombin III; Diagnostic Test: Protein C; Diagnostic Test: Protein S; Diagnostic Test: D-dimer; Diagnostic Test: Flow cytometry immunophenotyping
- control group: controlled group include healthy persons not suffering from acute leukemia either clinically or laboratory
  Interventions: Diagnostic Test: Antithrombin III; Diagnostic Test: Protein C; Diagnostic Test: Protein S; Diagnostic Test: D-dimer; Diagnostic Test: Flow cytometry immunophenotyping

INTERVENTIONS:
Diagnostic Test: Antithrombin III — quantitative measurement(%)
Diagnostic Test: Protein C — quantitative measurement(%)
Diagnostic Test: Protein S — quantitative measurement(%)
Diagnostic Test: D-dimer — quantitative measurement( ug/ml)
Diagnostic Test: Flow cytometry immunophenotyping — Flow cytometry immunophenotyping

SUMMARY:
The goal of this observational study is to evaluate the levels of Antithrombin III, Protein C, Protein S, and D-dimer in patients with Acute Leukemia (Acute Lymphoblastic Leukemia (ALL) and Acute Myeloid Leukemia (AML)). The main questions it aims to answer are:

What are the levels of Antithrombin III, Protein C, Protein S, and D-dimer in patients with Acute Lymphoblastic Leukemia? What are the levels of Antithrombin III, Protein C, Protein S, and D-dimer in patients with Acute Myeloid Leukemia? Researchers will compare patients with Acute Leukemia (30 with ALL and 30 with AML) to 30 healthy control subjects to see if there are significant differences in the levels of Antithrombin III, Protein C, Protein S, and D-dimer.

Participants will:

Undergo full history and clinical examination. Have routine hematological analysis including Complete Blood Count (CBC), blood film, Erythrocyte sedimentation rate (ESR), Prothrombin Time Test and INR (PT/INR), and partial thromboplastin time (PTT).

Have specific tests for quantitative measurement of Antithrombin III, Protein C, Protein S, and D-dimer.

Undergo Flow cytometry immunophenotyping.

ELIGIBILITY:
Inclusion Criteria:

1. patients with leukemia in group 1 and 2.
2. willing to participate in the study.

Exclusion Criteria:

1. refusing to participate.
2. patients with know to have either hereditary thrombophilia or current thrombosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will include 90 subjects, without regard to their sex or age. The subjects will be classified into two main groups: a patient group and a control group.
  Patient Group (Group 1): This group will consist of 60 patients suffering from acute leukemia. It is further divided into two subgroups:
  Group 1A: 30 patients diagnosed with acute lymphoblastic leukemia (ALL). Group 1B: 30 patients diagnosed with acute myeloid leukemia (AML). Patients will be selected from the outpatient clinic, internal medicine, and oncology departments at both Al Hussein and Sayed Galal University Hospitals, provided they give appropriate consent to participate.
  Control Group (Group 2): This group will consist of 30 healthy individuals who are not suffering from acute leukemia, as determined both clinically and through laboratory tests.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Antithrombin III, Protein C, Protein S, and D-dimer Levels in Acute Leukemia Patients | at the time of patient recruitment for the study.
  To evaluate and compare the quantitative levels of Antithrombin III, Protein C, Protein S, and D-dimer in patients diagnosed with Acute Lymphoblastic Leukemia (ALL) and Acute Myeloid Leukemia (AML) against healthy control subjects. This assessment will help determine any significant differences in these coagulation parameters within the different acute leukemia subtypes and in comparison to healthy individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Hussein University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) from this study, including de-identified demographic information, clinical examination findings, routine hematological analysis results (Complete Blood Count, Erythrocyte Sedimentation Rate, Prothrombin Time/INR, partial thromboplastin time), and specific test results (Antithrombin III, Protein C, Protein S, D-dimer, and Flow cytometry immunophenotyping), will be made available. The data will be provided in a secure, anonymized format suitable for secondary analysis (e.g., CSV or statistical software file types). This sharing aims to foster further research, facilitate meta-analyses, and enable validation studies by the wider scientific community, while strictly safeguarding participant privacy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified IPD will become available for access upon publication of the study's main results. The dataset will remain accessible for a period of ten (10) years following the initial publication date.
Access Criteria: Access to the IPD will be granted to qualified researchers for legitimate scientific purposes, subject to the following criteria:
  Submission of a detailed research proposal outlining the scientific objectives, methodology for analysis, and a commitment to ethical research practices.
  Approval of the research proposal by a designated Data Access Committee or institutional review board, if applicable, to ensure scientific merit and ethical considerations.
  Execution of a formal Data Use Agreement (DUA) with the study principal investigators, specifying the terms of data usage, confidentiality, data security, and a strict prohibition against any attempt at re-identification of participants.
  Agreement to acknowledge the original study and its investigators in any resulting publications or presentations.
  Confirmation that the proposed research aligns with the informed consent provided by study participants.